CLINICAL TRIAL: NCT04488523
Title: Leveraging Technology to Improve Family Relationships for Adolescents in Out-of-Home Placement
Brief Title: Family Telehealth Project for Foster Care Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Visa Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1928922
Record Dates: First submitted 2020-07-02; First posted 2020-07-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Parent-Child Relations; Communication
Keywords: telehealth; parent-child relationships; adolescent; Quality communication; Housing stability; Child welfare; Emotional regulation
MeSH Terms: conditions — Communication; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study is designed to iteratively adapt a family-based intervention with feedback from youth and caregiver participants and stakeholder partners, as well as to evaluate the feasibility, acceptability, and preliminary effectiveness of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-based Telehealth Treatment (Experimental): A family-based telehealth intervention.
  Interventions: Behavioral: Family-based Telehealth Intervention

INTERVENTIONS:
Behavioral: Family-based Telehealth Intervention — The Family Telehealth intervention focuses on improving parent-child relationships and communication.
  For the dyadic version, the intervention involves eleven hours of intervention material; it includes motivational interviews, individual and joint sessions co-led by two separate clinicians. The sessions will be delivered on a weekly basis.
  For the caregiver-only version, the intervention involves six hours of intervention material; it includes a motivational interview and individual sessions led by a single clinician. The sessions will be delivered on a weekly basis.

SUMMARY:
The purpose of this research is to adapt and evaluate the efficacy of an existing family based intervention to be delivered via telehealth to child welfare-involved (CWI) youth and their caregiver of origin.

DETAILED DESCRIPTION:
The goal of this study is to adapt and evaluate the efficacy of an existing empirically supported, family-based affect management intervention to be delivered via telehealth. There are two versions of this intervention: 1) a dyadic version to be delivered to CWI youth and their caregiver of origin, and 2) a caregiver-only version to be delivered to any caregiver (including kinship caregivers) of a CWI youth. The study involves iteratively adapting the intervention with feedback from youth and caregiver participants and stakeholder partners, as well as evaluating the feasibility, acceptability, and preliminary effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Eligible youth:

* Will be between the ages of 12 and 18 years
* Will have ongoing child welfare involvement
* Will be proficient in English
* Will have no cognitive impairment which would preclude provision of informed assent

Eligible caregivers for dyadic version:

* Will be the caregiver of origin for the enrolled youth
* Will be proficient in English or Spanish
* Will be cognitively capable of providing informed consent for themselves and their youth

Eligible caregivers for caregiver-only version:

* Will be the caregiver of a youth, between the ages of 12 and 18 years, with ongoing child welfare involvement
* Will be proficient in English or Spanish
* Will have no cognitive impairment which would preclude provision of informed consent

Exclusion Criteria:

* Caregivers whose rights were terminated due to substantiated abuse or neglect.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale | Immediately after the intervention.
  To measure caregiver and youth affect management skills. Scores range from 36 to 180, with higher scores indicating greater problems with emotion regulation.
Difficulties in Emotion Regulation Scale | Three months post-intervention.
  To measure caregiver and youth affect management skills. Scores range from 36 to 180, with higher scores indicating greater problems with emotion regulation.
Parent-adolescent General Communication Scale (PPAC) | Immediately after the intervention.
  To measure caregiver-youth communication. The PPAC measures both positive and negative communication. Scores for positive communication ranging from 7 to 35, with higher scores indicating more positive communication. Scores for negative communication range from 13 to 65, with higher scores indicating more negative communication.
Parent-adolescent General Communication Scale | Three months post-intervention.
  To measure caregiver-youth communication. The PPAC measures both positive and negative communication. Scores for positive communication ranging from 7 to 35, with higher scores indicating more positive communication. Scores for negative communication range from 13 to 65, with higher scores indicating more negative communication.

SECONDARY OUTCOMES:
Telehealth Satisfaction Questionnaire | Immediately after the intervention.
  To measure attitudes about the delivery of the intervention via telehealth.
Family telehealth feedback form | Two weeks post-baseline.
  To measure attitudes about the content and delivery of the intervention.
Family telehealth feedback form | Three weeks post-baseline.
  To measure attitudes about the content and delivery of the intervention.
Family telehealth feedback form | Four weeks post-baseline.
  To measure attitudes about the content and delivery of the intervention.
Family telehealth feedback form | Five weeks post-baseline.
  To measure attitudes about the content and delivery of the intervention.
Family telehealth feedback form | Nine weeks post-baseline.
  To measure attitudes about the content and delivery of the intervention.

OTHER OUTCOMES:
Family Assessment Device | Immediately after the intervention
  To measure general family functioning, affective responsiveness, and affective involvement. Scores range from 1 to 4 for each of the scales, with higher scores reflecting unhealthy family functioning.
Family Assessment Device | Three months post-intervention.
  To measure general family functioning, affective responsiveness, and affective involvement. Scores range from 1 to 4 for each of the scales, with higher scores reflecting unhealthy family functioning.
Stress Index for Parents of Adolescents | Immediately after the intervention.
  To measure caregiver-youth relationship quality and caregiver parenting stress. The items are scored on a 5-point rating scale, with raw scores then categorized as within normal limits, borderline, clinically significant, or clinically severe.
Stress Index for Parents of Adolescents | Three months post-intervention.
  To measure caregiver-youth relationship quality and caregiver parenting stress. The items are scored on a 5-point rating scale, with raw scores then categorized as within normal limits, borderline, clinically significant, or clinically severe.
Pediatric Symptom Checklist | Immediately after the intervention.
  To measure youth psychiatric symptoms. Scores range from 0 to 70, with scores of 30 or higher indicating psychological impairment.
Pediatric Symptom Checklist | Three months post-intervention.
  To measure youth psychiatric symptoms. Scores range from 0 to 70, with scores of 30 or higher indicating psychological impairment.
Homelessness Asset and Risk Screening Tool | Immediately after the intervention.
  To measure risk for homelessness and residential stability.
Homelessness Asset and Risk Screening Tool | Three months post-intervention.
  To measure risk for homelessness and residential stability.
Adolescent Risk Behavior Assessment | Immediately after the intervention.
  To measure youth substance use and youth sexual risk behavior.
Adolescent Risk Behavior Assessment | Three months post-intervention.
  To measure youth substance use and youth sexual risk behavior.
National Stressful Events Survey PTSD Short Scale | Immediately after the intervention.
  To assess the severity of posttraumatic stress disorder in youth. The item are scored on a 5-point rating scale (from 0 to 4). Scores range from 0 to 28, with higher scores indicating greater severity of acute stress disorder.
National Stressful Events Survey PTSD Short Scale | Three months post-intervention.
  To assess the severity of posttraumatic stress disorder in youth. The item are scored on a 5-point rating scale (from 0 to 4). Scores range from 0 to 28, with higher scores indicating greater severity of acute stress disorder.
Texas Christian University Drug Screen 5 - Opioid Supplement | Immediately after the intervention.
  To measure youth substance use.
Texas Christian University Drug Screen 5 - Opioid Supplement | Three months post-intervention.
  To measure youth substance use.
Asian American Family Conflict Scale | Immediately after the intervention.
  To assess caregiver perceptions of intergenerational acculturation conflict. The items are scored on a 5-point rating scale. Scores range from 10 to 50, with higher scores indicating greater family conflict.
Asian American Family Conflict Scale | Three months post-intervention.
  To assess caregiver perceptions of intergenerational acculturation conflict. The items are scored on a 5-point rating scale. Scores range from 10 to 50, with higher scores indicating greater family conflict.
DSM-5 Cross Cutting Symptom Inventory | Immediately after the intervention.
  To assess caregiver mental health domains that are important across psychiatric diagnoses. The items are scored on a 5-point rating scale (from 0 to 4). The score on each item within a domain should be reviewed. A rating of mild (i.e., 2) or greater on any item within a domain (except for substance use, suicidal ideation, and psychosis) and a rating of slight (i.e., 1) or greater on any item within a substance use, suicidal ideation, or psychosis domain may serve as a guide for additional inquiry and follow up to determine if a more detailed assessment for that domain is necessary.
DSM-5 Cross Cutting Symptom Inventory | Three months post-intervention.
  To assess caregiver mental health domains that are important across psychiatric diagnoses. The items are scored on a 5-point rating scale (from 0 to 4). The score on each item within a domain should be reviewed. A rating of mild (i.e., 2) or greater on any item within a domain (except for substance use, suicidal ideation, and psychosis) and a rating of slight (i.e., 1) or greater on any item within a substance use, suicidal ideation, or psychosis domain may serve as a guide for additional inquiry and follow up to determine if a more detailed assessment for that domain is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Folk JB, Valencia-Ayala C, Holloway ED, Anvar S, Czopp A, Tolou-Shams M. Feasibility and Acceptability of a Family-Based Telehealth Intervention for Families Impacted by the Child Welfare System: Formative Mixed Methods Evaluation. JMIR Form Res. 2024 Oct 15;8:e57939. doi: 10.2196/57939. PMID 39405104